CLINICAL TRIAL: NCT06609031
Title: Endoscopic Mucosal Resection Versus Cold Snare Polypectomy in the Treatment of Sessile Serrated Lesions Less Than 10mm in Size: a Single-center, Open-label, Randomized Controlled Trial
Brief Title: EMR Versus CSP in the Treatment of Sessile Serrated Lesions Less Than 10mm in Size
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024K225
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Sessile Serrated Lesion
Keywords: Sessile Serrated Lesion; cold snare polypectomy; endoscopic mucosal resection
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMR in treating SSLs less than 10mm in size (Experimental): The EMR procedure included the following: (1) needle injection of normal saline into the submucosa; (2) entrapment of the mucosal protrusion with a snare; and (3) resection using electrocautery
  Interventions: Procedure: endoscopic mucosal resection
- CSP in treating SSLs less than 10mm in size (Active Comparator): The CSP procedure included the following: (1) entrapment and resection of the polyp with a snare without electrocautery.
  Interventions: Procedure: Cold snare polypectomy

INTERVENTIONS:
Procedure: endoscopic mucosal resection — The SSLs less than 10mm in size in this group will be treated by EMR
  Arms: EMR in treating SSLs less than 10mm in size
Procedure: Cold snare polypectomy — The SSLs less than 10mm in size in this group will be treated by CSP
  Arms: CSP in treating SSLs less than 10mm in size

SUMMARY:
A prospective, single-center, open-label, randomized controlled study to compare the effectiveness and safety of endoscopic mucosal resection (EMR) and cold snare polypectomy (CSP) in treating colorectal sessile serrated lesions (SSLs) less than 10mm in size.

DETAILED DESCRIPTION:
1. Patients are undergone screening, surveillance, or therapeutic colonoscopy at the Endoscopy department of Gastrointestinal endoscopy center of Huadong hospital affiliated to Fudan University.
2. Randomize patients with suspicious sessile serrated lesions (SSLs) less than 10mm in size into 2 interventional groups based on Random function of Statistical Package for the Social Sciences (SPSS) 20.0, including (1) Group 1: Endoscopic mucosal resection (EMR) and (2) Group 2: Cold snare polypectomy (CSP).
3. Collecting variables which consist of primary and secodary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 35 and 75 years
* Suspected sessile serrated lesions less than 10mm in size in screening, surveillance or therapeutic colonoscopy
* 0-Is or 0-IIa according to Paris classification
* Type 1 according to NICE and JNET classification
* Type II according to pit pattern
* Patients must sign an informed consent form prior to registration in study

Exclusion Criteria:

* Unsuitable for removal by EMR or CSP
* Suspected dysplasia or malignancy
* Recurrent sessile serrated lesions after endoscopic resection
* Familial adenomatous polyposis, Lynch syndrome or serrated polyposis syndrome
* History of inflammatory bowel disease
* Patients taking anticoagulant and antiplatelet agents before the examination
* Severe illness or other high-risk conditions that prevent the patient from cooperating with or tolerating endoscopic therapy
* Refusal to sign the informed consent form or any other factors that are not suitable for enrollment or affect the ability to participate in the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
R0 resection | 2 weeks after the procedure
  Rate of R0 resection in treating SSLs less than 10mm in size

SECONDARY OUTCOMES:
en bloc resection | immediately after the procedure
  Rate of en bloc resection rate in treating SSLs less than 10mm in size
Vertical margins | 2 weeks after the procedure
  Rate of negative vertical margins in resected specimen
Lateral margin | 2 weeks after the procedure
  Rate of negative lateral margin in resected specimen
Presence of muscularis mucosae | 2 weeks after the procedure
  Rate of presence of muscularis mucosae in resected specimen
Presence of submucosa | 2 weeks after the procedure
  Rate of presence of submucosa in resected specimen
Clinically Significant Immediate Post-polypectomy Bleeding（CSIPB） | immediately after the procedure
  CSIPB was defined as any bleeding not responding to water jet irrigation or STSC and therefore requiring either coagu lation forceps or mechanical clips to achieve hemostasis
Clinically Significant Delayed Post-polypectomy Bleeding（CSDPB） | 2 weeks after the procedure
  CSPEB was defined as any bleeding after completion of the procedure requiring emergency room presentation, hospital isation or re-intervention (endoscopy, angiography, surgery).
Delayed perforation | 2 weeks after the procedure
  Rate of delayed perforation in treating SSLs less than 10mm in size

CONTACTS AND LOCATIONS:
Overall Officials: Danian Ji, M.D., Study Director — Huadong Hospital
Locations (1):
- Huadong hospital affiliated to Fudan university, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)